CLINICAL TRIAL: NCT00098202
Title: Randomized Placebo-Controlled Trial (RPCT) of Maize/Zinc in Guatemala
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); Fogarty International Center of the National Institute of Health (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Cancer Institute (NCI) (NIH); RTI International (Other); University of Colorado, Denver (Other); Center for Studies of Sensory Impairment, Aging and Metabolism (Other); Foundation for Alimentation and Nutrition, Central America and Panama (Other); USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: GN 06; U01HD040657 (NIH)
Record Dates: First submitted 2004-12-03; First posted 2004-12-06 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Nutrition; Pregnancy
Keywords: Global Network; Micronutrients; Zinc; Maternal and child health; Women's health; International; Guatemala; Nutrition; Corn; Maize
MeSH Terms: conditions — Callosities | interventions — Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Low phytic acid maize
Drug: Zinc

SUMMARY:
Malnutrition is a serious health problem in the developing world. This study looks at the effects of changing the type of basic food staple (corn) used in Guatemala and infant zinc supplementation on infants' growth, development, and illnesses from infectious diseases.

DETAILED DESCRIPTION:
Poor mineral nutrition, especially deficiencies of iron and zinc, is a major cause of maternal and, especially, infant morbidity/mortality in developing world countries. The objectives of this study are to determine whether: a) linear growth velocity between 6 and 12 months in infants receiving a 5mg Zn supplement will be greater than that for infants receiving placebo; b) linear growth velocity will be greater for infants receiving complementary foods containing low phytate maize than for the infants fed wild-type control maize. In addition, Zn metabolic studies will be performed. The objective of the metabolic studies are to measure key variables of Zn homeostasis in maternal participants during changes in the reproductive cycle and in infants during a time when they are most vulnerable to Zn deficiency.

The primary outcome measurement is linear growth velocity between 6 and 12 months. Secondary outcomes are weight gain, diarrheal incidence/prevalence and infant neurodevelopmental measures. Optional maternal and infant biochemical data will be collected from a convenience sample comprised of willing participants.

One additional component to this study is to collect information on the nutritional status of the women receiving low-phytate vs. control maize and the infants enrolled in this study.

The current protocol for infants in this study specifies measurements of exchangeable zinc pool (EZP) at 6 and 12 months of age; in order to lessen the burden of study participation we plan to conduct the metabolic studies in infants at only nine months of age. In addition to decreasing the number of infant studies, this change will enable families who are only participating in the metabolic studies (not simultaneously enrolled in the sibling cohort) to cease all study demands at the end of the nine month measurement (an overall decrease of three months in study participation).

The primary outcome measure for this study is the quantity of zinc absorbed (mg/day)from complementary foods and a Zn supplement at age 9 months. The rationale for measures of zinc absorption in infants is that the low phytate complementary feeding is expected to have a beneficial public health effect only if it results in enhanced mineral, especially zinc, absorption. Therefore, confirmation of increased zinc absorption can be regarded as the first logical stage of any efficacy study.

The sample size of 420 is required in order to observe a 6% increase in growth rates for Zn supplemented infants compared to placebo treated infants within each maize group with 80% power.

ELIGIBILITY:
Inclusion criteria:

* Informed consent of mother
* Mother between the ages of 18 and 40 years
* Mother typically eats homemade tortillas
* Mother typically eats a minimum of 15 homemade tortillas per day.
* Mother resides in a community served by the Comalapa, Chimaltenango, Community Health Center in the Western Highlands of Guatemala

Exclusion criteria:

* Other member of the dwelling unti already enrolled in the study.
* Mother has more than eight living children.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 420 (Estimated)
Dates: Start 2003-03; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Infant Maize/Zn Supplementation Trial:
Linear growth velocity
Zn Homeostasis Studies:
Measures of zinc homeostasis

SECONDARY OUTCOMES:
Infant Maize/Zn Supplementation Trial:
Weight gain
Morbidity
Infant neurodevelopment
Maternal and infant biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hambidge, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Community, Comalapa, Guatemala

REFERENCES:
- [Derived] Hambidge KM, Mazariegos M, Kindem M, Wright LL, Cristobal-Perez C, Juarez-Garcia L, Westcott JE, Goco N, Krebs NF. Infant stunting is associated with short maternal stature. J Pediatr Gastroenterol Nutr. 2012 Jan;54(1):117-9. doi: 10.1097/MPG.0b013e3182331748. PMID 21866055
- See also: Global Network for Women's and Children's Health Research — http://gn.rti.org
- See also: Research Triangle Institute International — http://www.rti.org